CLINICAL TRIAL: NCT05461261
Title: A Randomized Controlled Trial to Evaluate the Efficacy and Safety of Docetaxel Combined With Platinum-based Drugs Compared With Docetaxel Alone for Metastatic Hormone-sensitive Prostate Cancer Patients Carrying DNA Repair Mutation
Brief Title: The Efficacy and Safety of Docetaxel Combined With Platinum for Metastatic Hormone-sensitive Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUNU-PC-114
Record Dates: First submitted 2022-07-13; First posted 2022-07-18 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Hormone Sensitive Metastatic Prostate Cancer; DNA Damage Repair Deficiency; Chemotherapy Effect; Chemotherapeutic Toxicity
MeSH Terms: interventions — Docetaxel; prednisolone acetate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Docetaxel plus platinum (Experimental): Docetaxel combined with platinum-based drugs will be applied every 3 weeks for 6 cycles.
  Interventions: Drug: Docetaxel; Drug: Prednisolone Acetate; Drug: Platinum-based drugs
- Docetaxel alone (Active Comparator): Docetaxel alone will be applied every 3 weeks for 6 cycles.
  Interventions: Drug: Docetaxel; Drug: Prednisolone Acetate

INTERVENTIONS:
Drug: Docetaxel — Docetaxel will be given intravenously 75 mg/m2 every 3 weeks for 6 cycles.
Drug: Prednisolone Acetate — 5mg Prednisolone Acetate will be given orally twice a day during treatment.
Drug: Platinum-based drugs — Platinum-based drugs will be given intravenously 70 mg/m2 every 3 weeks for 6 cycles. Cisplatin or carboplatin will be carefully chosen according to each patient's Creatinine Clearance.
  Arms: Docetaxel plus platinum

SUMMARY:
This randomized controlled trial was designed to evaluate the efficacy and safety of Docetaxel combined with Platinum-based drugs compared with Docetaxel alone for metastatic hormone-sensitive prostate cancer patients carrying DNA repair mutation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 40 and ≤75 years of age.
* All patients must have been histologically diagnozed of prostate cancer.
* Metastatic disease confirmed by imaging: positive bone scan, or soft tissue or visceral metastases confirmed by abdominal/pelvic/chest contrast CT or MRI or PSMA PET-CT scan.
* Participants who were treated with androgen deprivation therapy (ADT) (LHRH agonist/antagonist or orchectomy) with or without first-generation anti-androgens within 12 weeks prior to random assignment must maintain serum testosterone castration levels, i.e., ≤50 ng/dL (≤ 1.75 nmol/L) during the study period. First-generation anti-androgens must be discontinued at least 1 day before the start of study therapy.
* Participants must carry one of the following DNA repair gene mutation: 1) HRR-related genes: ATM, BARD1, BRCA1, BRCA2, BRIP1, CDK12, CHEK1, CHEK2, FANCL, PALB2, RAD51B, RAD51C, RAD51D, RAD54L; 2) Lynch syndrome-related genes: EPCAM, MLH1, MSH2, MSH6, PMS2.
* Eastern Cooperative Oncology Group (ECOG) physical condition score ≤1.
* Patients must have adequate hematologic function, hepatic function and renal function within 28 days prior to registration.
* Patients must participate voluntarily and sign an informed consent form(ICF), indicating that they understand the purpose and required procedures of the study, and are willing to participate in. Patients must be willing to obey the prohibitions and restrictions specified in the research protocol.
* Sexually active male subjects and their partner must agree the use of condoms as an effective contraceptive method and to avoid sperm donation during the whole treatment and within 4 weeks after the end of treatment.

Exclusion Criteria:

* Patients with neuroendocrine, small cell, or signet ring cell histological features are not eligible.
* Patients with brain/meningeal metastases are not eligible..
* Patients previously received any of the following treatments are not eligible: 1) LHRH agonists/antagonists within 12 weeks prior to the start of study therapy; 2) Second generation androgen receptor (AR) inhibitors, such as enzaluamine, dalotamide, apatamide, etc; 3) Cytochrome P17 enzyme inhibitors (e.g., abiraterone acetate or oral ketoconazole) as antitumor therapy for PCa; 4) Chemotherapy (including docetaxel) or immunotherapy for PCa; 5) Systemic corticosteroids > 10 mg/day equivalent dose of prednisone within 28 days prior to random assignment.
* Patients who were known to have hypersensitivity to any research drug or similar drug are not eligible.
* Patients received local treatments such as pre-focal treatment,radiotherapy and palliative endoscopic resection
* Patients with severe or uncontrolled concurrent infections are not eligible.
* Patients must not have New York Heart Association Class III or IV congestive heart failure at the time of screening. Patients must not have any thromboembolic event, unstable angina pectoris, myocardial infarction within 6 months prior to registration.
* Patients must not have uncontrolled severe hypertension, persistent uncontrolled diabetes, oxygen-dependent lung disease, chronic liver disease, or HIV infection.
* Patients must not have had other malignancies other than prostate cancer in the past 5 years, but cured basal cell or squamous cell skin cancers can be enrolled.
* Patients with mental illness, mental disability or inability to give informed consent are not eligible.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to Metastatic Castration-Resistant Prostate Cancer (mCRPC) | up to 3 years
  Time from treatment initiation to Metastatic Castration-Resistant Prostate Cancer (mCRPC). Patients with metastatic prostate cancer develop PCa progression during androgen deprivation therapy (or after bilateral orchiectomy), meet any of the following criteria was defined as mCRPC. 1)PSA progression (defined as elevated PSA levels(≥1ng/ml) for no less than 2 measurements at least 1 week apart); 2) Radiographic progression in soft tissues, with or without PSA progression, according to RECIST 1.1 criteria; 3) Bone progression (defined as 2 or more new bone lesions on bone scans) with or without PSA progression, according to PCWG.

SECONDARY OUTCOMES:
Overall survival | up to 5 years
  The survival rate of participants during follow-up time.
rPFS | up to 5 years
  Radiographic progression-free survival. The survival of participants without radiographic progression.
Time to PSA progression | up to 5 years
  PSA progression is defined as elevated PSA levels(≥2ng/ml) for no less than 2 measurements at least 1 week apart.
Time to subsequent anti-tumor therapy | up to 5 years
  Time from end of treatment to the time when subsequent anti-tumor therapy is needed.
Adverse events | up to 3 years
  All grades of adverse events will be recorded according to NCI CTCAE (v.5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Hongqian Guo, Study Chair — Nanjing Drum Tower Hospital, affiliated to medical school of Nanjing University Locations: China, Jiangsu
Locations (1):
- Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided